CLINICAL TRIAL: NCT00868907
Title: A Crossover Study to Assess the Relative BA of Delayed-release Risedronate Compared When Dosed With Either Dinner, Breakfast or Breakfast Plus a Calcium/Vitamin D Tablet
Brief Title: Study Assessing Dosing Time and Calcium and Vitamin D on the Relative BA of 35 mg DR Risedronate Dosed With Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008138
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
MeSH Terms: interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): 35 mg risedronate DR tablet administered within 5 minutes after completing a standard breakfast and taking one Caltrate® 600+D tablet
  Interventions: Drug: 35 mg risedronate DR tablet
- Treatment B (Experimental): 35 mg risedronate DR oral tablet administered within 5 minutes after completing a standard dinner
  Interventions: Drug: 35 mg risedronate DR tablet
- Treatment C (Active Comparator): 35 mg risedronate DR oral tablet administered within 5 minutes after completing a standard breakfast
  Interventions: Drug: 35 mg risedronate DR tablet

INTERVENTIONS:
Drug: 35 mg risedronate DR tablet — 35 mg risedronate DR oral tablet administered within 5 minutes after completing a standard breakfast and taking one Caltrate® 600+D tablet
  Arms: Treatment A
Drug: 35 mg risedronate DR tablet — 35 mg risedronate DR oral tablet administered within 5 minutes after completing a standard dinner
  Arms: Treatment B
Drug: 35 mg risedronate DR tablet — 35 mg risedronate DR oral tablet administered within 5 minutes after completing a standard breakfast
  Arms: Treatment C

SUMMARY:
Randomized, open-label, single dose, 3-treatment, 3-period crossover study, with a 14- to 17-day washout period between doses. The study will consist of a screening visit, study center admission (preceding Treatment Periods 1, 2 and 3), 3 treatment periods (4 days each), 1 washout period (14 to 17 days separating periods 1, 2 and 3), and exit procedures.

ELIGIBILITY:
Inclusion Criteria:

* female, 40 to 70 years of age
* non-lactating and either surgically sterile or postmenopausal
* body mass index less than or equal to 32 kg/m2 at screening

Exclusion Criteria:

* no use of a bisphosphonate within 1 month
* no history of GI disease
* no use of any medications within 7-14 days prior to scheduled dosing day

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Relative BA of DR Risedronate dosed: After breakfast and with calcium/vitamin D tablet, compared to DR Risedronate dosed after breakfast After dinner compared to DR Risedronate administered after breakfast. | 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Chantell Wilson, PhD, Study Director — Procter and Gamble
Locations (4):
- United States (4):
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Evansville, Indiana